CLINICAL TRIAL: NCT03592420
Title: Efficacy of a Multifactorial and Personalized Program for Fall Prevention in Community-dwelling Elderly in Comparison to the Usual Care: a Randomized Controlled Trial
Brief Title: PRE.C.I.S.A - Fall Prevention and Promotion of Active and Healthy Aging
Acronym: PRECISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Unita' Sanitaria Locale Di Modena (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Modena (Other); Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRUA2-2013-00002056
Record Dates: First submitted 2018-06-25; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Fall; Aging; Parkinson Disease; Stroke
Keywords: Accidental falls; Clinical trial; Aged; Parkinson's Disease; Stroke; Exercise; Education
MeSH Terms: conditions — Parkinson Disease; Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interdisciplinary interventions (Experimental): Multicomponent interventions
  * On-site supervised group exercise program (11 weeks)
  * Educational / behavioral sessions addressing specific behavioral and environmental risk factors for falls delivered by trained health professionals (11 sessions in total)
  * Home visits for suggestion and implementations of safety interventions aiming at reducing environmental hazards
  * Home-based exercise program: Personalized multi-factorial interventions: patients will have geriatric, neurology and physiatrist outpatient referrals to assess and treat individual risk factors.
  Personalized multi-factorial interventions. Patients will have geriatric, neurology and physiatrist outpatient referrals to assess and treat individual risk factors
  Interventions: Behavioral: Interdisciplinary multicomponent interventions
- Usual care (Active Comparator): Usual care: after pre-test assessment and randomization, participants in the control group will be given a structured booklet with detailed information about participant's own personal risk factors (fall risk profile) to be given to the family doctor, together with an information booklet on fall risk factors and their prevention.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Interdisciplinary multicomponent interventions
  Arms: Interdisciplinary interventions
Behavioral: Usual care — standard care
  Arms: Usual care

SUMMARY:
Randomized Controlled Trial (RCT) aiming at assessing the efficacy of an interdisciplinary multi-component and personalized multi-factorial intervention for reducing falls at one year post-enrolment in comparison to the usual care in a sample of community dwelling elderly (age ≥65 years), with or without Parkinson's Disease and/or previous Stroke.

DETAILED DESCRIPTION:
BACKGROUND: Current literature on fall prevention for community-dwelling elderly who are at risk of falling suggests that: 1) either single, multicomponent or multifactorial interventions are effective at preventing falls; 2) elderly at risk of falling with Parkinson's Disease (PD) and previous Stroke, although having an even greater risk of falling, are often excluded by these interventions; 3) often, present screening methods for risk of falling do not allow the early identification of subjects at risk before the first fall.

AIMS

* To compare the efficacy of an interdisciplinary multicomponent and personalized multifactorial intervention aiming at reducing falls in comparison to the usual care, in a sample of community dwelling elderly, with or without Parkinson's Disease and/or previous Stroke, within the context of an RCT.
* To improve the accuracy of screening tests for risk of falling by using wearable inertial sensors.
* To develop a reduced set of clinical and instrumental indicators, to be utilized as a quick and reliable screening tests in outpatients clinics.

METHODS: multicenter, randomized controller trial, with blind assessments on pretest, postest and on one-year follow-up.

POPULATION: community-dwelling elderly (aged ≥65 years) with age-related or neurological condition-related (Parkinson's Disease and/or Stroke) risk of falling.

INTERVENTION: interdisciplinary multi-component (group-based exercise; home-based exercise; increasing knowledge/education; home safety interventions) and personalized multi-factorial interventions (assessment and treatment of individual fall risk factors) CONTROL: structured information about participant's own personal risk factors given to the family doctor.

OUTCOMES: The primary endpoint is the fall rate at one year in both groups. The secondary endpoint is the fall risk at one year.

EXPECTED RESULTS: in the intervention group, a significant reduction in the number of total fall is expected, together with decreases indicators of utilization of acute health services because of falls. At three months, it is expected a significant improvement of functioning (motor functions, activity and participation) and health quality indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling elderly (aged ≥65 years)
2. Moderate to high fall risk, either associated to aging or to neurological diseases as Parkinson's Disease and stroke.
3. Ability to walk 10 meters without assistance (walking aid permitted)
4. Informed consent to participation

Exclusion Criteria:

1. Whatever concurrent medical condition which may constitutes a contraindication to physical exercise
2. Known cognitive decline or an established diagnosis of dementia (mini mental score >24) or an evident cognitive decline on pre-enrolment which would be likely to impair the ability of comprehension of simple instructions and / or of collaborating
3. Severe hearing impairment, so that a subject will not understand less than 80% of ordinary conversation with/or without hearing aids.
4. Severe hypovision, not counteracted by lenses, which will limit the patient in executing at least one activity of daily living (for instance, necessity of assistance for walking because of visual deficit).
5. Severe aphasia or visuo-spatial deficits, to the extent that these impairments will limit significantly the ability to comprehend (orally or visually) simple instructions.
6. Acute vertigo or dizziness lasting less than 3 months
7. Regular participation to other exercise program that it is likely to challenge balance, including physical therapy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 366 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Fall rate at 12 months from enrolment | Months 1 - Months 12
  The primary endpoint will be the total number of falls (fall rate) occurred in each arm within 12 months from enrolment. This endpoint will be recorded by participants in a fall diary (which will be collected from each participant at month 12). Recorded information in the fall diary will be monitored monthly with follow-up calls

SECONDARY OUTCOMES:
Risk of falling at 12 months from enrolment | Months 1 - Months 12
  This secondary endpoint will be calculated as the number of patients with at least one falls within 12 months from enrolment. This endpoint will be recorded by participants in a fall diary (which will be collected from each participant at month 12). Recorded information in the fall diary will be monitored monthly with follow-up calls
Percentage of falls associated to hospital admission at 12 months from enrolment | Months 1 - Months 12
  This secondary endpoint will be recorded by participants in a fall diary (which will be collected from each participant at month 12). Recorded information in the fall diary will be monitored monthly with follow-up calls
Severity of the fall | Months 1 - Months 12
  This secondary endpoint will be recorded by participants in a fall diary (which will be collected from each participant at month 12). Recorded information in the fall diary will be monitored monthly with follow-up calls
Mortality attributable to fall | Months 1 - Months 12
  This secondary endpoint will be recorded by participants in a fall diary (which will be collected from each participant at month 12). Recorded information in the fall diary will be monitored monthly with follow-up calls
Fall-free interval time | Months 1 - Months 12
  This secondary endpoint will be recorded by participants in a fall diary (which will be collected from each participant at month 12). Recorded information in the fall diary will be monitored monthly with follow-up calls
Total number of A&E accesses attributable to falls | Months 1 - Months 12
  This secondary endpoint will be recorded by participants in a fall diary (which will be collected from each participant at month 12). Recorded information in the fall diary will be monitored monthly with follow-up calls
Risk of A&E access attributable to falls | Months 1 - Months 12
  This secondary endpoint will be recorded by participants in a fall diary (which will be collected from each participant at month 12). Recorded information in the fall diary will be monitored monthly with follow-up calls
Length of stay as inpatient attributable to falls | Months 1 - Months 12
  This secondary endpoint will be recorded by participants in a fall diary (which will be collected from each participant at month 12). Recorded information in the fall diary will be monitored monthly with follow-up calls

CONTACTS AND LOCATIONS:
Overall Officials: Fabio La Porta, MD, Principal Investigator — AZIENDA USL DI MODENA
Locations (2):
- Italy (2):
  - Nuovo Ospedale Civile Sant'Agostino Estense, Modena
  - Arcispedale "Santa Maria Nuova" di Reggio Emilia, Reggio Emilia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gillespie LD, Robertson MC, Gillespie WJ, Sherrington C, Gates S, Clemson LM, Lamb SE. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007146. doi: 10.1002/14651858.CD007146.pub3. PMID 22972103
- [Result] Weiss A, Herman T, Plotnik M, Brozgol M, Giladi N, Hausdorff JM. An instrumented timed up and go: the added value of an accelerometer for identifying fall risk in idiopathic fallers. Physiol Meas. 2011 Dec;32(12):2003-18. doi: 10.1088/0967-3334/32/12/009. Epub 2011 Nov 17. PMID 22094550
- [Result] Schoene D, Wu SM, Mikolaizak AS, Menant JC, Smith ST, Delbaere K, Lord SR. Discriminative ability and predictive validity of the timed up and go test in identifying older people who fall: systematic review and meta-analysis. J Am Geriatr Soc. 2013 Feb;61(2):202-8. doi: 10.1111/jgs.12106. Epub 2013 Jan 25. PMID 23350947
- [Derived] La Porta F, Lullini G, Caselli S, Valzania F, Mussi C, Tedeschi C, Pioli G, Bondavalli M, Bertolotti M, Banchelli F, D'Amico R, Vicini R, Puglisi S, Clerici PV, Chiari L; PRECISA Group. Efficacy of a multiple-component and multifactorial personalized fall prevention program in a mixed population of community-dwelling older adults with stroke, Parkinson's Disease, or frailty compared to usual care: The PRE.C.I.S.A. randomized controlled trial. Front Neurol. 2022 Sep 1;13:943918. doi: 10.3389/fneur.2022.943918. eCollection 2022. PMID 36119666